CLINICAL TRIAL: NCT04977037
Title: Feasibility and Effectiveness of Home-based Telerehabilitation Program for Recovery of Upper Limb Functions in Incomplete Spinal Cord Injury
Brief Title: A Telerehabilitation Program for SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Mission Connect a project of TIRR Foundation (Unknown)
Responsible Party: Principal Investigator, Nuray Yozbatiran, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-21-0114
Record Dates: First submitted 2021-06-25; First posted 2021-07-26 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: Cervical Spinal Cord Injury; upper limb; tDCS; telerehabilitation

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: active or sham tDCS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Experimental): Anodal transcranial direct current stimulation (tDCS) targeting the primary motor cortex delivered at 2mA for 20 minutes
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): Sham transcranial direct current stimulation (tDCS) targeting the primary motor cortex delivered at 2mA for 20 minutes
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Anodal tDCS will be placed over the primary motor cortex and delivered at 2mA for 20 minutes. Immediately after stimulation ceases, participants will continue with unilateral repetitive arm and finger exercises for 60 minutes. Exercise difficulty will gradually be increased and adjusted per participant's tolerance.
  Arms: Active tDCS
Device: Sham tDCS — Anodal tDCS will be placed over the primary motor cortex and delivered at 2mA for 20 minutes. Immediately after stimulation ceases, participants will continue with unilateral repetitive arm and finger exercises for 60 minutes. Exercise difficulty will gradually be increased and adjusted per participant's tolerance.
  Arms: Sham tDCS

SUMMARY:
This study evaluates a remotely supervised, home-based therapeutic program to improve upper-limb voluntary movement in adults with tetraplegia caused by incomplete spinal cord injury (iSCI).

DETAILED DESCRIPTION:
Spinal Cord Injury (SCI) has been associated with serious reduction in functional independence. Despite compelling evidence that treatment intensity has a profound effect on motor recovery only a small fraction of SCI population are able to receive intensive in-clinic treatment. Difficulty traveling to the clinic, poor adherence to assignments and high cost are limiting factors. Currently, telerehabilitation programs are emerging as an alternative effective method of delivery for rehabilitation services. The literature and our preliminary findings support the model that augmentation of activity in spared corticospinal tract (CST) axons is a critical mechanism of motor improvement, and furthermore that CST activity can be increased by repetitive motor training and by electrical stimulation of the primary motor cortex (M1). However, there is still lack of knowledge on safety, feasibility and efficacy of remotely- supervised home-based therapy programs that incorporates non-invasive brain stimulation and high intensity repetitive arm exercises. To address these questions, 36 adults (above 18 years) with cervical SCI will be randomly assigned to two groups in a 2:1 ratio (active stimulation group, n=24 vs control group, n=12) and receive daily treatment, 10 sessions, over 2-weeks. The anodal tDCS will be applied over primary motor cortex (M1) at an intensity of 2mA for 20 minutes and proceed with 60 minutes of repetitive arm and hand training. Primary outcome measure is change in Graded and Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) from baseline to immediately after treatment and 4-weeks follow-up. The session will be supervised in real-time via videoconferencing.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of a chronic incomplete cervical lesion as defined by the American Spinal Injury Association Impairment scale classification and at least for 6 months post-injury;
2. upper-extremity weakness associated with tetraplegia with minimal residual thumb and index; finger movement sufficient to grip small objects such as marble;
3. no brain injury;
4. no planned alteration in upper-extremity therapy or medication for muscle tone during the course of the study;
5. no contradiction to tDCS;
6. access to internet at home.

Exclusion Criteria:

1. prior history of seizure;
2. chronic use of neuroactive medication (e.g., neurostimulants, anticonvulsants, or antidepressants);
3. any joint contracture or severe spasticity in the affected upper extremity, as measured by a Modified Ashworth Score ≥ than 3 out of 4.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nuray Yozbatiran, PhD, PT, Principal Investigator — The University of Texas Health Sciences Center at Houston
Locations (1):
- The Institute for Rehabilitation and Research (TIRR) at Memorial Hermann, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 13 | 7
Completed | 11 | 6
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (16.5) | 45.8 (12.1) | 46.2 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 10 | 3 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 7 | 20
Asia Impairment Scale Classification [Count of Participants; unit: Participants] — The Asia Impairment Scale (AIS) categorizes spinal cord injury severity based on sensory and motor function loss.
  AIS Classification:
  A = Complete: No motor/sensory function in the sacral segments S4-S5 B = Incomplete: Sensory but not motor function below the neurological level, includes the sacral segments S4-S5 C = Incomplete: Below the neurological level, motor function preserved and more than 50% of key muscles have a muscle grade < 3 D = Incomplete: Below the neurological level, motor function persevered and at least 50% of key muscles have a muscle grade ≥3
  Participants
    A | 0 | 0 | 0
    B | 5 | 2 | 7
    C | 1 | 5 | 6
    D | 7 | 0 | 7
Time Since Injury [Mean (Standard Deviation); unit: Months] | 84 (104.2) | 71 (85.12) | 79.89 (96.41)

OUTCOME MEASURES:

1. Primary Outcome: Arm and Hand Function as Assessed by Score on the Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP)
Description: The Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) assesses the integration of sensorimotor hand and upper limb impairment and function. GRASSP total score will be reported, and it ranges from 0 to 116, with a higher score indicating a higher level of arm and hand function.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
score on a scale | 64.9 (25.5) | 58.3 (31.1)

2. Primary Outcome: Arm and Hand Function as Assessed by Score on the Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP)
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
score on a scale | 68 (28.8) | 59.7 (32.6)

3. Primary Outcome: Arm and Hand Function as Assessed by Score on the Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 6
score on a scale | 72.1 (28.3) | 57.7 (37.7)

4. Secondary Outcome: Adherence With the Therapy as Assessed by the Number of Sessions Participants Attended
Time Frame: Treatment Day 1- Day 10
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
sessions | 9.6 (0.65) | 9.0 (1.73)

5. Secondary Outcome: Adherence With the Therapy as Assessed by the Number of Participant Drop-outs
Time Frame: Between enrollment and 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
Participants | 2 | 1

6. Secondary Outcome: Feasibility of Home Intervention as Indicated by Participants' Perceptions of Usefulness of the Intervention as Assessed by the Visual Analog Scale (VAS)
Description: Participants rated the usefulness of the interventions on a scale of 0 to 10, with 0 indicating not useful at all and 10 indicating very useful.
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
score on a scale | 9.1 (1.3) | 9.1 (0.9)

7. Secondary Outcome: Grip Strength
Description: Maximum force generated by hand muscles and measured with a hand-held dynamometer
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
pounds (lbs) | 19.2 (25.6) | 9.3 (7.5)

8. Secondary Outcome: Grip Strength
Description: Maximum force generated by hand muscles and measured with a hand-held dynamometer
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
pounds (lbs) | 20.9 (25.7) | 10.8 (10.1)

9. Secondary Outcome: Grip Strength
Description: Maximum force generated by hand muscles and measured with a hand-held dynamometer
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 6
pounds (lbs) | 24.6 (31.5) | 11.3 (10.7)

10. Secondary Outcome: Self Care as Assessed by Score on the Self Care Subscale of the Spinal Cord Injury Independence Measure (SCIM III)
Description: Total score on the Self Care Subscale of the Spinal Cord Injury Independence Measure (SCIM III) ranges between 0 to 20, with a higher score indicating a higher level of independence in daily functions.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
score on a scale | 11.1 (6.4) | 6.4 (5.8)

11. Secondary Outcome: Self Care as Assessed by Score on the Self Care Subscale of the Spinal Cord Injury Independence Measure (SCIM III)
Description: as for outcome 10
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
score on a scale | 11.5 (6.1) | 7.3 (6.4)

12. Secondary Outcome: Self Care as Assessed by Score on the Self Care Subscale of the Spinal Cord Injury Independence Measure (SCIM III)
Description: as for outcome 10
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 6
score on a scale | 11.6 (6.1) | 7.5 (5.8)

13. Secondary Outcome: Number of Participants Who Had Adverse Events
Time Frame: from baseline to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
Participants | 1 | 2

14. Secondary Outcome: Feasibility of Home Intervention as Indicated by Participants' Perceptions of Level of Difficulty of Using tDCS as Assessed by the Visual Analog Scale (VAS)
Description: Participants rated the level of difficulty of using tDCS on a scale of 0 to 10, with 0 indicating not difficult at all and 10 indicating very difficult
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
score on a scale | 1.1 (1.3) | 1 (1.1)

15. Secondary Outcome: Feasibility of Home Intervention as Indicated by Participants' Perceptions of Level of Difficulty of Using Exercise Equipment as Assessed by the Visual Analog Scale (VAS)
Description: Participants rated the level of difficulty of using exercise equipment on a scale of 0 to 10, with 0 indicating not difficult at all and 10 indicating very difficult.
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 7
score on a scale | 1.1 (1.3) | 1.7 (1.5)

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7
Other Adverse Events (participants affected / at risk) | 1/13 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS (N=13) | Sham tDCS (N=7)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 0 | 1
Autonomic Dysreflexia (AD) (Nervous system disorders) | 0 | 1
Pelvic pain on right side (Musculoskeletal and connective tissue disorders) | 0 | 1
Sick day during home therapy (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT04977037/Prot_SAP_000.pdf